CLINICAL TRIAL: NCT03634085
Title: A Single Ascending Dose Trial Investigating the Safety, Tolerability and Pharmacokinetics of Orally Administered BDM-2 in Healthy Male Subjects
Brief Title: Single Ascending Dose Trial Investigating Safety, Tolerability and Pharmacokinetics of BDM-2 in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hivih (Industry)
Collaborators: Venn Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BDM-2-C001
Record Dates: First submitted 2018-08-02; First posted 2018-08-16 (Actual); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: safety; tolerability; pharmacokinetics
MeSH Terms: interventions — Suspensions

STUDY DESIGN:
Intervention Model Description: In Sessions I to VI, 6 single, orally administered ascending doses of BDM-2 or placebo will be investigated, alternately dosed in 2 cohorts of 8 healthy male subjects each (Cohorts A and B). For each dose, 6 subjects will receive active treatment and 2 subjects will receive placebo. Subjects will be randomized in such a way that for each dose different subjects receive placebo. In Sessions I to VI, doses are planned to be administered under fasted conditions.
Who Masked: Participant, Investigator
Masking Description: double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Ascending doses of BDM-2 in Bottle (50 mg - 3600 mg); oral suspension or placebo will be orally administered and will be investigated, alternately dosed in Cohort A of 8 healthy male subjects under fasted conditions. For each dose, 6 subjects will receive active treatment and 2 subjects will receive placebo. Subjects will be randomized in such a way that for each dose different subjects receive placebo.
  The last session for the subjects in Cohort A will be under fed conditions where the same treatment allocation as in the session of the selected dose (administered under fasted conditions) will be used.
  Interventions: Drug: BDM-2 in Bottle (50 mg - 3600 mg); oral suspension
- Cohort B (Experimental): Ascending doses of BDM-2 in Bottle (50 mg - 3600 mg); oral suspension or placebo will be orally administered and will be investigated, alternately dosed in Cohort B of 8 healthy male subjects under fasted conditions. For each dose, 6 subjects will receive active treatment and 2 subjects will receive placebo. Subjects will be randomized in such a way that for each dose different subjects receive placebo.
  Interventions: Drug: BDM-2 in Bottle (50 mg - 3600 mg); oral suspension

INTERVENTIONS:
Drug: BDM-2 in Bottle (50 mg - 3600 mg); oral suspension — BDM-2 in bottle will be reconstituted with a 100 mL vehicle (0.2% Sodium Dodecyl Sulfate and water) to achieve a suspension for oral administration.

SUMMARY:
This is a first-in-human (FIH), double-blind, placebo-controlled, randomized trial in healthy adult male subjects, to evaluate the safety, tolerability and pharmacokinetics (PK) of single ascending oral doses of BDM-2. The effect of food on the PK of a single dose of BDM-2 will also be evaluated.

DETAILED DESCRIPTION:
The Sponsor HIVIH is developing a new antiretroviral medicine, BDM-2, for the potential treatment of Human Immunodeficiency Virus (HIV). The study will investigate the safety, tolerability and pharmacokinetics (PK) (how well the medicine is taken up by the body) of single doses of the test medicine given by mouth, in healthy male volunteers. The effect of food on the PK of the test medicine will also be assessed.

This is the first time the medicine will be dosed in humans. Over 6 study periods, ascending (increasing) doses of the test medicine or placebo (dummy drug) will be given to 16 healthy male volunteers in the fasted state. Alternately dosed to two groups each made up of 8 volunteers. After each dose volunteers will remain in the clinical unit for 48 hours for blood samples to be taken and safety assessments to be performed.

To investigate the effect of food, it is planned that in Period 7 the medicine will be administered in the fed state. On the 7th study period one of the doses administered in a previous period will be administered under fed conditions (with food). Each volunteer will receive 3 or 4 single doses of test medicine or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male aged between 18 and 55 years at screening, inclusive.
2. Body Mass Index (BMI) 18.0-32.0 kg/m2 at screening, inclusive.
3. Good physical and mental health as established by medical history, physical examination, respiratory rate, electrocardiogram (ECG) and vital signs (including body temperature) recording, and results of biochemistry, coagulation, hematology and urinalysis tests during screening as judged by the investigator.
4. Non-smoker/non-user of nicotine containing products for at least 3 months prior to screening, to be confirmed by a urine cotinine dipstick test at screening and on Day -1 of the first session.
5. Availability and willingness to complete the trial and follow the instructions of the investigator or trial-site personnel.
6. Willing and able to adhere to the prohibitions and restrictions specified in the protocol
7. Easy venous accessibility.
8. Must have signed an Informed Consent Form (ICF) prior to screening, indicating that he understands the purpose of, and procedures required for the trial, and is willing to participate in the trial.
9. Must agree to provide a blood sample for DNA research.
10. Subject who is heterosexually active with a woman of childbearing potential must agree to use 2 effective methods of birth control (i.e., male condom with either female intrauterine device, diaphragm, cervical cap or hormone-based contraceptive), during the trial and for at least 90 days after receiving the last dose of trial medication. If the female sexual partner is postmenopausal for at least 2 years, or is surgically sterile (has had a total hysterectomy, bilateral oophorectomy, or bilateral tubal ligation/bilateral tubal clips without reversal operation), or otherwise is incapable of becoming pregnant, the birth control methods mentioned are not applicable, however, subjects should use a condom during the trial and for at least 90 days after receiving the last dose of trial medication to prevent unintended exposure via the ejaculate.

    Subjects who had vasectomy and have a female partner of childbearing potential must use a male condom during the trial and for at least 90 days after receiving the last dose of trial medication.

    Note: A male and female condom should not be used together due to risk of breakage or damage caused by latex friction.

    Note: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial medication (during the trial and for at least 90 days after receiving the last dose of trial medication). The reliability of sexual abstinence needs to be evaluated in relation to the duration of the trial and the preferred and usual lifestyle of the subject.

    Note: Subjects will be instructed that if their partner becomes pregnant during the trial this should be reported to the investigator. The investigator should also be notified of pregnancy occurring during the trial but confirmed after completion of the trial. In the event that a subject's partner is subsequently found to be pregnant after the subject is included in the trial, then consent will be sought from the partner and, if granted, any pregnancy will be followed and the status of mother and/or child will be reported to the sponsor after delivery.
11. Must agree not to donate sperm during the trial and for at least 90 days after receiving the last dose of trial medication.

Exclusion Criteria:

1. History of or current clinically significant medical illness including (but not limited to) gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, endocrinologic, genitourinary, renal, hepatic, respiratory, inflammatory, neoplastic, or infectious disease, or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the trial results.
2. Clinically significant abnormalities of hematology or biochemistry (out of range values should be considered as to their significance and the subject not included if the value is considered to be detrimental). This includes but is not limited to liver function tests.
3. Subjects with Gilbert's syndrome.
4. Clinically significant presence or history of allergy or intolerance (including lactose), or presence or history of clinically significant allergy requiring treatment, as judged by the investigator (hay fever is allowed unless it is active).
5. Positive serology for hepatitis A virus (HAV) immunoglobulin M (IgM), hepatitis B virus surface antigen (HBsAg), anti-hepatitis C virus antibodies (anti-HCV-AB), or anti HIV antibodies 1+2 (anti-HIV-AB 1+2) at screening.
6. History of alcohol or drug abuse within the last 2 years before screening or positive test result(s) for alcohol and/or drugs of abuse at screening or on Day -1 of first session.
7. Regular alcohol consumption >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
8. Surgery of gastro-intestinal tract that might interfere with absorption (subjects who have had cholecystectomy may be included). Subject has currently significant and active diarrhea, nausea, or constipation that in the investigator's opinion could influence drug absorption or bioavailability.
9. Intake of any disallowed therapies before the first dose of trial medication (on Day 1 of the first session).
10. Donation of blood or blood products or substantial loss of blood (more than 500 mL) within 3 months before first dose of trial medication (on Day 1 of the first session) or the intention to donate blood or blood products during the trial
11. Major surgery, fracture, or prolonged immobilization (more than 2 weeks) within 3 months preceding screening, or surgery has been planned during the time the subject is expected to participate in the trial.
12. Unable to swallow solid, oral dosage forms (multiple capsules) whole with the aid of water (subjects may not chew, divide, dissolve, or crush the trial medication).
13. Plans to father a child while enrolled in the trial or within 90 days after receiving the last dose of trial medication.
14. History of hypersensitivity or idiosyncrasy to any of the components of the investigational drug.
15. Participation in a clinical trial within 3 months before first dose of trial medication (on Day 1 of the first session).
16. Participation in a trial of an investigational product or an experimental medical device within 3 months or within a period less than 5 times the drug's half-life, whichever is longer, prior to the first dose (on Day 1 of the first session) or during this trial.
17. Trial site employee or immediate family members of a trial site or sponsor employee.
18. Have previously been enrolled in this trial.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MB ChB, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

REFERENCES:
- [Derived] Bonnard D, Le Rouzic E, Singer MR, Yu Z, Le Strat F, Batisse C, Batisse J, Amadori C, Chasset S, Pye VE, Emiliani S, Ledoussal B, Ruff M, Moreau F, Cherepanov P, Benarous R. Biological and Structural Analyses of New Potent Allosteric Inhibitors of HIV-1 Integrase. Antimicrob Agents Chemother. 2023 Jul 18;67(7):e0046223. doi: 10.1128/aac.00462-23. Epub 2023 Jun 13. PMID 37310224

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Ascending doses of BDM-2 in Bottle (50 mg - 3600 mg); oral suspension or placebo will be orally administered and will be investigated, alternately dosed in Cohort A of 8 healthy male subjects under fasted conditions. For each dose, 6 subjects will receive active treatment and 2 subjects will receive placebo. Subjects will be randomized in such a way that for each dose different subjects receive placebo.
  The last session for the subjects in Cohort A will be under fed conditions where the same treatment allocation as in the session of the selected dose (administered under fasted conditions) will be used.
  BDM-2 in Bottle (50 mg - 3600 mg); oral suspension: BDM-2 in bottle will be reconstituted with a 100 mL vehicle (0.2% Sodium Dodecyl Sulfate and water) to achieve a suspension for oral administration.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 8 | 8
Period 1 | 8 (8 subjects started BDM2-50 mg and 8 subjects completed BDM2-50 mg including matching placebo.) | 8 (8 subjects started BDM2 - 150mg and 8 subjects completed BDM2 - 150 mg including matching placebo)
Period 2 | 8 (8 subjects started BDM2 - 450 mg and 7 subjects completed BDM2 - 450 mg (drop out; 1 active)) | 8 (8 subjects started BDM2 - 900 mg fasted and 8 subjects completed BDM2 - 900 mg fasted)
Period 3 | 8 (8 subjects started BDM2 - 1800 mg and 7 subjects completed BDM2 - 1800 mg (drop out; 1 active)) | 8 (8 subjects started and 6 subjects completed BDM2 - 900 mg fed (dropout; 1 active 1 placebo))
Period 4 | 8 (8 subjects started BDM2 - 3100 mg and 7 subjects completed BDM2 - 3100 mg (drop out; 1 active)) | 0 (this period is not applicable for Cohort B)
Completed | 7 (1 subject dropped out due to car accident) | 6 (1 subject dropped out due to personal emergency 1 subject dropped out due to personal circumstances)
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (9.8) | 36.6 (10.4) | 34.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Related Adverse Event, Including Abnormal Laboratory Events
Description: All AEs, including clinical laboratory, vitals signs, body temperature, respiratory rate, physical examinations and ECGs will be analyzed in all subjects receiving BDM-2.
Time Frame: up to 4 months
Population: The same 8 subjects attended Period 1-4 for Cohort A and 8 other subjects attended Period 1-3 for Cohort B, therefore all randomized subjects who received at least 1 dose of trial medication are displayed in this section. For both cohorts this are 8 subjects, so all AEs per cohort are based on 8 subjects.
Measure: Number; unit: participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 8 | 8
participants
  placebo: number analyzed (Participants) | 8 | 5
  placebo | 1 | 3
  50 mg CohA - 150mg Coh B: number analyzed (Participants) | 5 | 6
  50 mg CohA - 150mg Coh B | 2 | 4
  450mg CohA - 900mg fast CohB: number analyzed (Participants) | 6 | 6
  450mg CohA - 900mg fast CohB | 4 | 9
  1800mg CohA - 900mg fed CohB: number analyzed (Participants) | 5 | 5
  1800mg CohA - 900mg fed CohB | 4 | 4
  3100mg Coh A: number analyzed (Participants) | 5 | 0
  3100mg Coh A | 3 |

ADVERSE EVENTS:
Time Frame: 4 months
Description: Each cohort has 8 subjects. Cohort A subjects attended Period 1-4 and Cohort B subjects attended Period 1-3.
  Arm A has 4 interventions in 8 subjects (6 on active, 2 on placebo) and Arm B has 3 intreventions in 8 subjects (6 on active and 2 on placebo).
  The affected subjects in Cohort A cannot be more than 8 subjects and the same accounts for Cohort B.
  There were a couple of dropouts, therefore the amount of affected subjects differs in placebos and other arms between the interventions.
Groups:
- Cohort A-placebo; Cohort A-50mg; Cohort A-450mg; Cohort A-1800mg; Cohort A-3100mg: Ascending doses of BDM-2 in Bottle (50 mg - 3600 mg); oral suspension or placebo will be orally administered and will be investigated, alternately dosed in Cohort A of 8 healthy male subjects under fasted conditions. For each dose, 6 subjects will receive active treatment and 2 subjects will receive placebo. Subjects will be randomized in such a way that for each dose different subjects receive placebo.
  The last session for the subjects in Cohort A will be under fed conditions where the same treatment allocation as in the session of the selected dose (administered under fasted conditions) will be used.
  BDM-2 in Bottle (50 mg - 3600 mg); oral suspension: BDM-2 in bottle will be reconstituted with a 100 mL vehicle (0.2% Sodium Dodecyl Sulfate and water) to achieve a suspension for oral administration.
- Cohort B-placebo; Cohort B-150mg; Cohort B-900mg Fasted; Cohort B-900mg Fed: Ascending doses of BDM-2 in Bottle (50 mg - 3600 mg); oral suspension or placebo will be orally administered and will be investigated, alternately dosed in Cohort B of 8 healthy male subjects under fasted conditions. For each dose, 6 subjects will receive active treatment and 2 subjects will receive placebo. Subjects will be randomized in such a way that for each dose different subjects receive placebo.
  BDM-2 in Bottle (50 mg - 3600 mg); oral suspension: BDM-2 in bottle will be reconstituted with a 100 mL vehicle (0.2% Sodium Dodecyl Sulfate and water) to achieve a suspension for oral administration.
Arm/Group | Cohort A-placebo | Cohort B-placebo | Cohort A-50mg | Cohort B-150mg | Cohort A-450mg | Cohort B-900mg Fasted | Cohort A-1800mg | Cohort B-900mg Fed | Cohort A-3100mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/5 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/8 | 2/5 | 2/5 | 3/6 | 2/6 | 5/6 | 4/5 | 2/5 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A-placebo (N=8) | Cohort B-placebo (N=5) | Cohort A-50mg (N=5) | Cohort B-150mg (N=6) | Cohort A-450mg (N=6) | Cohort B-900mg Fasted (N=6) | Cohort A-1800mg (N=5) | Cohort B-900mg Fed (N=5) | Cohort A-3100mg (N=5)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Dysgeusia
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Abdominal pain upper
Abdomonal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Abdominal mass
loss of contiousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — loss of contiousness
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — muscle spasma
arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — arthropod bite
skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — skin abrasion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall have no right to publish the Research Output, without the Customer's prior written consent. The Parties make their best efforts to reach an agreement on the issue of conditions of the publication of the Reseach Output. In case of repeated disagreement, Customer shall be the sole Party to decide in its capacity of Sponsor under what conditions and release period the Research Output should be published.

DOCUMENTS (3):
  • Study Protocol (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT03634085/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT03634085/SAP_001.pdf
  • Informed Consent Form (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT03634085/ICF_002.pdf